CLINICAL TRIAL: NCT03753763
Title: 12-weeks, Multicentre, Randomized, Double-blind, Placebo-controlled, Exploratory, Pilot Study to Evaluate the Safety and Efficacy of Safinamide 200 mg OD, as add-on Therapy, in Patients With Possible or Probable Parkinsonian Variant of MSA
Brief Title: Safinamide for Multiple System Atrophy (MSA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z7219K01; 2018-004145-16 (EudraCT Number)
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-07

CONDITIONS: Multiple System Atrophy
Keywords: MSA, safinamide
MeSH Terms: conditions — Multiple System Atrophy; Thyroid Dyshormonogenesis 2A | interventions — safinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Safinamide methanesulfonate film-coated tablets once daily
  Interventions: Drug: Safinamide Methanesulfonate
- Placebo (Placebo Comparator): Safinamide Methanesulfonate matching placebo film-coated tablets once daily
  Interventions: Drug: Safinamide Methanesulfonate matching placebo

INTERVENTIONS:
Drug: Safinamide Methanesulfonate — 100 mg (free base)
  Other Names: Xadago
  Arms: Active
Drug: Safinamide Methanesulfonate matching placebo — 100 mg placebo
  Other Names: placebo
  Arms: Placebo

SUMMARY:
The study is a placebo controlled study, with two parallel arms, in which participants will be randomly assigned in a 2:1 ratio to receive either active (200 mg safinamide) or placebo in a double blind manner. Study population is patients diagnosed, with possible or probable parkinsonian variant of Multiple System Atrophy who are on a stable treatment of levodopa

DETAILED DESCRIPTION:
The overall design is a parallel group, placebo controlled, double blind study. The target population are participants diagnosed with possible or probable parkinsonian variant of Multiple System Atrophy who are on stable doses of levodopa.

Trial participation will be up to a maximum duration of 14 weeks and will comprise a screening period (up to 2 weeks), a 2-week run in period during which subjects will receive 1 tablet (either 100 mg safinamide or matching placebo), followed by a 10-week period, during which study participants will take 2 tablets of study medication (200 mg safinamide or placebo) once daily, taken in the morning in addition to their morning levodopa dose. A telephone follow-up call will be performed 2 weeks after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 30 to 80 years of age inclusive, at the time of signing the informed consent;
2. Participants who are diagnosed (with MRI confirmation) with possible or probable parkinsonian variant of Multiple System Atrophy less than 2 years ago;
3. Participants with an anticipated survival of at least 3 years in the opinion of the investigator;
4. Female not pregnant, not breastfeeding, and at least one of the following conditions applies:

   * Not a woman of childbearing potential OR
   * A woman of childbearing potential who agrees to follow the contraceptive guidance during the treatment period and for at least 30 days after the last dose of study intervention;
5. Capable of giving signed informed consent

Exclusion Criteria:

1. History of neurosurgical procedure, including stereotactic surgery;
2. History of Deep Brain Stimulation (DBS);
3. History of bipolar disorder, severe depression, schizophrenia or other psychotic disorder;
4. History of drug and/or alcohol abuse within 12 months prior to screening as defined by the current edition of the Diagnostic and Statistical Manual of Mental Disorders;
5. History of dementia (DSM-V criteria);
6. Ophthalmologic history including any of the following conditions: albinism, uveitis, retinitis pigmentosa, retinal degeneration, active retinopathy, severe progressive diabetic retinopathy, inherited retinopathy or family history of hereditary retinal disease;
7. Active hepatitis B or C;
8. History of human immunodeficiency virus (HIV) infection;
9. Subjects not able to swallow oral medications;
10. Subjects with severe orthostatic symptoms;
11. Impaired ambulation, i.e. falling more than once per week, bedridden patients or confined to a wheelchair during the whole day;
12. Subjects with active malignant neoplasms;
13. Movement disorders other than MSA (e.g. Parkinson Disease, dementia with Lewy bodies, essential tremor, progressive supranuclear palsy, pharmacological or post-encephalic parkinsonism);
14. Any clinically significant or unstable medical or surgical condition that, in the opinion of the investigator, might preclude safe completion of the study or might affect the results of the study;
15. Not on a stable regime, for at least 4 weeks prior to the randomization (baseline visit), of

    1. oral levodopa (including controlled release, immediate release or a combination of controlled release/immediate release), with or without benserazide/carbidopa, with or without addition of a catechol O-methyltransferase (COMT) inhibitor or
    2. dopamine agonist, anticholinergic and/or amantadine.
16. Patients should not have received treatment with monoamine oxidase inhibitors in the 2 weeks prior to the randomization visit, nor treatment with levodopa infusion, pethidine, opiates, opioids, fluoxetine, fluvoxamine in the 4 weeks prior to the randomization visit;
17. Patients should not have received treatment with an oral or depot neuroleptic within 12 weeks prior to the randomization visit;
18. Use of any investigational drug within 30 days prior to screening or 5 half-lives, whichever is the longest;
19. Montreal Cognitive Assessment (MoCA) ≤ 20;
20. Laboratory assessments showing moderate or severe hepatic impairment (2x ULN);
21. Allergy/sensitivity or contraindications to the investigational medicinal products (IMPs) or their excipients, anticonvulsants, levodopa or other anti-parkinsonian drugs;
22. Any clinically significant condition which, in the opinion of the Investigator, would not be compatible with study participation or represent a risk for patients while in the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Keywood, MD, Study Director — Zambon SpA
Locations (19):
- Italy (11):
  - Università di Bologna, Bologna
  - AAST degli Spedali Civili di Brescia, Brescia
  - San Raffaele Cassino, Cassino
  - Fondazione Università "G. D'Annunzio", Chieti
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedaliera Universitaria - Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Opsedaliero Universitaria Pisana, Pisa
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Universitaria OO.RR. San Giovanni di Dio - Ruggi d'Aragona, Salerno
  - Azienda Ospedaliera Santa Maria di Terni, Terni
- Spain (8):
  - Hospital General Universitario de Elche, Alicante
  - Hospital de Cruces, Barakaldo
  - Hospital de la Santa Creu i Sant Pau Barcelona, Barcelona
  - Hospital Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen de Rocio, Seville

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 56 participants were planned to be screened in order to achieve 49 participants randomly assigned (2:1) to study drug and 42 evaluable participants, resulting in a planned estimated total of 32 evaluable participants receiving safinamide and 17 evaluable participants receiving matching placebo. Only 42 completed the study while 7 discontinued it.
Pre-assignment Details: Participants (males and females between 30 and 80 years) diagnosed with possible or probable parkinsonian variant of MSA <2 years before, with MRI consistent with the diagnosis of MSA, and not suggesting an alternative explanation to the clinical diagnosis of MSA, and with an anticipated survival of at least 3 years in the opinion of the Investigator.
Groups:
- Safinamide: Safinamide methanesulfonate film-coated tablets once daily. During the titration period of 2 weeks (Week 1 to Week 2) participants received 1 tablet (100 mg) safinamide, while during the treatment period (Week 3 to Week 12) they received 2 tablets (200 mg) safinamide once-a-day, taken in the morning, in addition to their daily levodopa dose.
- Placebo: Safinamide methanesulfonate matching placebo film-coated tablets once daily. Safinamide matching placebo was administered both during the titration period of 2 weeks (Week 1 to Week 2) and during the following period (Week 3 to Week 12), once daily, taken in the morning, in addition to their daily levodopa dose.
Period: Overall Study
Arm/Group | Safinamide | Placebo
Started | 32 | 17
Completed (Completed the study (at week 14)) | 26 | 16
Not Completed | 6 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — clinical deterioration | 1 | 0

BASELINE CHARACTERISTICS:
Population: The ITT Population included all randomized participants. This population was used for describing all the demographic characteristics and all efficacy variables.
Groups:
- Total: Total of all reporting groups
Arm/Group | Safinamide | Placebo | Total
Number analyzed (Participants) | 32 | 17 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 11 | 28
  >=65 years | 15 | 6 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (8.23) | 62.8 (10.27) | 64.7 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 6 | 26
  Male | 12 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 31 | 17 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 23 | 13 | 36
  Spain | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: TEAEs (Treatment Emergent Adverse Events) and SAEs (Serious Adverse Events)
Description: While evaluating safety and tolerability of safinamide, 200 mg od, compared with placebo, severity of TEAEs, their relationship to study drug, their seriousness and their consequences were assessed. TEAEs were defined as adverse events (AEs) that started after the first dose of study drug.
Time Frame: Throughout the study, from baseline (and at each interim visit) to telephone follow-up visit at 14 week.
Population: The Safety Population included all randomized participants who took at least 1 dose of study drug. This population was used to summarize all safety data.
Measure: Number; unit: events
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 32 | 17
events
  Any TEAEs | 52 | 28
  Mild TEAEs | 49 | 21
  Moderate TEAEs | 4 | 5
  Severe TEAEs | 3 | 4
  Serious TEAEs | 2 | 0
  Study drug-related TEAEs | 15 | 11
  TEAEs leading to study drug withdrawal | 1 | 0
  AEs leading to death | 1 | 0

2. Secondary Outcome: Change From Baseline to Week 12 in the Goniometric Measurement for Anterior Displacement
Description: To evaluate the potential efficacy of safinamide 200 mg od, as add-on therapy, on quality of life (change in anterior displacement). The goniometric measurement consists in the posture evaluation of the patient, measuring through a goniometer the angle of the flexion of the trunk. Goniometric measurement of "anterior" displacement was determined using a wall goniometer and expressing the value in degrees in the range of 0 to 90.
Time Frame: From baseline to week 12
Population: The ITT Population included all randomized participants. This population was used for all efficacy variables.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 32 | 17
degrees | 1.3 (9.46) | 0.9 (8.01)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; The model included treatment, week of visit, and treatment-by-visit interaction as fixed effects and baseline score as a covariate; Test type: Superiority; p = 0.9697, Mixed Models Analysis; A mixed-model repeated measures (MMRM) was used to analyze the change in anterior and lateral displacement from baseline; Least square mean difference = 0.1, 95% CI 2-sided [-6.3 to 6.5]

3. Secondary Outcome: Change From Baseline to Week 12 in the Goniometric Measurement for Lateral Displacement
Description: To evaluate the potential efficacy of safinamide 200 mg od, as add-on therapy, on quality of life (change in anterior displacement). The goniometric measurement consists in the posture evaluation of the patient, measuring through a goniometer the angle of the flexion of the trunk. Goniometric measurement of "lateral" displacement was determined using a wall goniometer and expressing the value in degrees in the range of 0 to 90.
Time Frame: From baseline to week 12
Population: The ITT Population included all randomized participants. This population was used for all efficacy variables.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 32 | 17
degrees | 1.3 (5.08) | -0.2 (4.47)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.7751, Mixed Models Analysis — A mixed-model repeated measures (MMRM) was used to analyze the change in anterior and lateral displacement from baseline; least square mean difference = 0.5, 95% CI 2-sided [-3.1 to 4.1]

4. Secondary Outcome: Change From Baseline to Week 12 in Unified Multiple System Atrophy Rating Scale (UMSARS), Part II (ITT Population)
Description: UMSARS is a validated, disease-specific scale representing the diverse signs and symptoms in MSA. Higher scores on the UMSARS scales mean poorer health.
  UMSARS has the following domains:
  Part I - Activities of Daily Living score (12 questions ranged in 0-4 [total score 0-48]) that evaluates motor including autonomic activities Part II - Motor Examination score (14 questions, [total score 0-56]) Part III - Autonomic Examination Part IV - Global disability scale ((1=completely independent; 2=not completely independent; 3=more dependent; 4=very dependent; 5=total dependent and helpless).
  Only UMSARS Part II total score is reported, which was obtained as the sum of the 14 items in the scale. If any of the items were missing, then the total score was considered missing. Higher scores indicate worse functional situation.
Time Frame: From baseline to week 12
Population: The ITT Population included all randomized participants. This population was used for all efficacy variables.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 32 | 17
score on a scale | -0.1 (5.40) | -0.4 (5.85)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.9076, Mixed Models Analysis; A mixed-model repeated measures (MMRM) was used to analyze the change in from baseline in UMSARS Part II; least square mean difference = 0.2, 95% CI 2-sided [-3.3 to 3.7]

5. Secondary Outcome: Change From Baseline to Week 12 in Unified Multiple System Atrophy Rating Scale (UMSARS), Part II (PP Population)
Description: as for outcome 4
Time Frame: From baseline to week 12
Population: The Per Protocol Population will include all randomized participants who do not have any entry criteria violations or protocol deviations that could significantly impact the assessment or interpretation of efficacy data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 21 | 13
score on a scale | -1.1 (4.66) | -0.6 (6.17)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.5386, Mixed Models Analysis; A mixed-model repeated measures (MMRM) was used to analyze the change in from baseline in UMSARS Part II; least square mean difference = -1.1, 95% CI 2-sided [-4.8 to 2.6]

6. Secondary Outcome: Change From Baseline to Week 12 in Multiple System Atrophy Health-Related Quality of Life (MSA-QoL) Scale
Description: The MSA-QoL is a self-reported questionnaire focusing on MSA-specific symptoms and has a scale ranging from 0 to 160, with 0= 'no problem' and 160= "extreme problem".
Time Frame: From baseline to week 12
Population: The ITT Population included all randomized participants. This population was used for all efficacy variables
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 32 | 17
units on a scale | 5.6 (25.57) | -2.9 (14.37)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3364, Mixed Models Analysis; A mixed-model repeated measures (MMRM) was used to analyze the change in from baseline in MSA-QoL scale; Least square mean difference = 6, 95% CI 2-sided [-6.5 to 18.6]

7. Secondary Outcome: Change From Baseline to Week 12 in Montreal Cognitive Assessment (MoCA) Scale
Description: The Montreal Cognitive Assessment (MoCA) was designed as a tool for rapid screening for mild cognitive impairment. It evaluates different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructive skills, abstraction, calculation and orientation. The administration time of the MoCa is 10 minutes. The MoCA scale ranges from 0 to 30, with higher scores indicating better cognitive functioning.
Time Frame: From baseline to week 12
Population: The ITT Population included all randomized participants. This population was used for all efficacy variables.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 32 | 17
score on a scale | 0.0 (2.01) | -0.3 (2.09)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; The ANCOVA included change from baseline as the response variable, treatment group as a factor, and baseline score as a covariate; Test type: Superiority; p = 0.7574, ANCOVA; Least square mean difference = 0.2, 95% CI 2-sided [-1.1 to 1.5]

8. Secondary Outcome: Change From Baseline to Week 12 in Unified Dystonia Rating Scale (UDRS)
Description: UDRS consists of a Historical Section, divided into questionnaires about 1) on-dyskinesia and 2) off -dystonia, and an Objective Section, divided into 3) impairment and 4) disability scales. The Historical Section is scored from 0-60, and the Objective section is scored 0-44, where higher scores reflect greater difficulty or impairment.
  The Unified Dystonia Rating Scale (UDRS) assesses the motor severity and duration of dystonia in 14 body areas. The total score, obtained as the sum of the severity and duration factors, ranges from 0 to 112. Higher scores indicate worse dystonia.
Time Frame: From baseline to week 12
Population: The ITT Population included all randomized participants. This population was used for all efficacy variables.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Safinamide | Placebo
Number analyzed (Participants) | 32 | 17
units on a scale | 1.0 (4.82) | 0.3 (5.60)
Statistical Analysis 1: Comparison: Safinamide vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.6393, Mixed Models Analysis; A mixed-model repeated measures (MMRM) was used to analyze the change from baseline in UDRS; Least square mean difference = 0.8, 95% CI 2-sided [-2.5 to 4.0]

ADVERSE EVENTS:
Time Frame: At baseline, at interim visits (Weeks 2 - 8, and more precisely at days 14 ± 3, 28 ± 3, 56 ± 3), at End of Treatment visit (EOT) at Week 12 (84 ± 3 days), and at follow-up call at week 14 ( 98 ± 3).
Arm/Group | Safinamide | Placebo
All-Cause Mortality (participants affected / at risk) | 1/32 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/32 | 0/17
Other Adverse Events (participants affected / at risk) | 21/32 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safinamide (N=32) | Placebo (N=17)
Cardiac respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safinamide (N=32) | Placebo (N=17)
Asthenia (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (7) | 5 (5)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Parkinsonian gait (Nervous system disorders) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 2 (4)
Dependent rubor (Vascular disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT03753763/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT03753763/SAP_001.pdf